CLINICAL TRIAL: NCT00759252
Title: Perceptions Regarding Investigational Screening for Memory Problems in Primary Care: The PRISM-PC Study
Brief Title: Perceptions Regarding Investigational Screening for Memory Problems in Primary Care
Acronym: PRISM-PC
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Malaz Boustani, MD, MPH, Regenstrief Institute, IU Center for Aging Research Scientist, Indiana University
Other Study IDs: IA0141; R01AG029884 (NIH); 5R01AG029884-02 (NIH)
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Dementia
Keywords: diagnosis of dementia; perceptions of risk; dementia screening
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to conduct a cross-sectional survey of primary care patients to better understand their perceptions of the risks and benefits of a screen and subsequent diagnostic confirmation of dementia.

DETAILED DESCRIPTION:
The Health Belief Model was used to explore the public's acceptance or enthusiasm for early recognition of dementia. Based on this model, prior research and clinical experiences, and a systematic literature review, the PRISM-PC instrument was developed. The PRISM-PC items seek to capture both the patient's acceptance of dementia screening and the patient's perception of potential harms and benefits of such screening. The instrument includes questions regarding screening by performance-based questionnaires, blood tests, or brain imaging.

The PRISM-PC instrument includes 50 items that are organized into 8 sets of questions that cover the following areas:

A) Prior experience with AD (5 items) B) Acceptance of screening for AD (6 items) C) Acceptance of screening for other conditions (2 items) D) Benefits of screening for AD (9 items) E) Stigma of screening for AD (10 items) F) Impact of screening for AD on independence (6 items) G) Suffering of screening for AD (4 items) H) Demographics (7 items) Excluding section A and H (prior experience with AD and demographics), each item of the six other sections is rated on a 5-point Likert scale (strongly agree, agree, don't know, disagree, and strongly disagree).

Based on the previous PRISM-PC pilot study (a survey response rate of 80%) and the Dementia screening and diagnosis study (screening acceptance rate of 90%, positive dementia screening rate of 20% among participants aged 70 and older, and dementia diagnostic acceptance rate of 50%), a total of 1,500 volunteers will be approached. A random selection of 200 participants will be re-administered the questionnaire within one week to test the short-term temporal stability of their responses (test-retest).

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and older
* At least one office visit to their primary care physician within the last year
* No chart-based diagnosis of dementia or memory problem
* Willing to sign a consent form to participate in the study

Exclusion Criteria:

* Does not speak English
* Too hearing-impaired to hear the informed consent statement or the survey
* Severe mental illness based on the patient's electronic medical charts

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 954 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Primary care patients' perceptions of the risks and benefits of early identification of dementia | Measurement will continue through the duration of the study

SECONDARY OUTCOMES:
Evaluation of the association between primary care patients' acceptance for early identification of dementia and their perceptions of the risks and benefits of such identification after adjusting for potential confounders such as demographics | Measurement will continue through the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Malaz Boustani, MD, MPH, Principal Investigator — Regenstrief Institute, Center for Aging Research
Locations (1):
- Indiana University Medical Group, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Schubert CC, Boustani M, Callahan CM, Perkins AJ, Hui S, Hendrie HC. Acute care utilization by dementia caregivers within urban primary care practices. J Gen Intern Med. 2008 Nov;23(11):1736-40. doi: 10.1007/s11606-008-0711-0. Epub 2008 Aug 9. PMID 18690489
- [Background] Boustani M, Perkins AJ, Monahan P, Fox C, Watson L, Hopkins J, Fultz B, Hui S, Unverzagt FW, Callahan CM, Hendrie HC. Measuring primary care patients' attitudes about dementia screening. Int J Geriatr Psychiatry. 2008 Aug;23(8):812-20. doi: 10.1002/gps.1983. PMID 18232061
- [Background] Brayne C, Fox C, Boustani M. Dementia screening in primary care: is it time? JAMA. 2007 Nov 28;298(20):2409-11. doi: 10.1001/jama.298.20.2409. No abstract available. PMID 18042918